CLINICAL TRIAL: NCT06458452
Title: Enhancing Immersion in Virtual Reality Based Advanced Life Support Training Through Artificial Intelligence Driven Voice Control: A Randomized Controlled Trial
Brief Title: Enhancing Immersion in Virtual Reality Based Advanced Life Support Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Dilek Kitapçıoğlu, Assist Prof Dr, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Acibadem CASE
Record Dates: First submitted 2024-06-03; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Advanced Cardiac Life Support; Artificial Intelligence
Keywords: Virtual Reality; Advanced Cardiac Life Support; Artificial Intelligence; Voice Recognition; Serious Gaming
MeSH Terms: interventions — Advanced Cardiac Life Support

STUDY DESIGN:
Who Masked: Participant
Masking Description: Fourth semester students of Vocational School of Anaesthesiology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game Interaction with Voice Recognition (Group VG) (Active Comparator): Group VG participants will use AI driven Voice Recognition as game controller interface.
  Interventions: Other: Using Virtual Reality based serious gaming module for Advanced Cardiac Life Support
- Game Interaction with VR Controllers (Group CG) (Active Comparator): Group CG participants will use hand held VR controllers as game controller interface.
  Interventions: Other: Using Virtual Reality based serious gaming module for Advanced Cardiac Life Support

INTERVENTIONS:
Other: Using Virtual Reality based serious gaming module for Advanced Cardiac Life Support — Group VG will use Artificial Intelligence driven Voice Recognition as an interface for game control whereas Group CG will only use hand held Virtual Reality controllers as an interface for game control

SUMMARY:
Virtual Reality based training modulues have become a part of simulation based medical education and are nowadays used for undergraduate and postgraduate level training of healthcare professionals.In parallel to the advancements in Artificial Intelligence technology voice regotnition has the potential to be used as an interfeace during game play .The aim of this study is whether game interface with Artificial Intelligence based voice regognition may elevate the level of immersion during the use of Virtual Reality based serious gaming for Advanced Cardiac Life Support Training.

DETAILED DESCRIPTION:
Virtual Reality based training modules have become one of the training modalities for simulation based healthcare training and have an important role for the training of healthcare professionals VR based training modules have used hand-held controllers for navigation and interaction with the virtual environment so far. In parallel to the advancements in Artificial Intelligence (AI) and natural language processing (NLP) potential for voice command interfaces, offer an alternative method of control in Virtual Reality applications by providing more intuitive and accessible means of interaction for users.Voice commands, powered by NLP algorithms, enable users to navigate and manipulate virtual environments using natural language and have the potential to reduce the learning curve associated with Virtual Reality controller inputs. Voice interfaces have also the potential to offer accessibility benefits for users with physical disabilities, for whom conventional controllers may be difficult to use].

Despite the potential advantages, using voice command systems in Virtual Reality gaming has also its limitations like speech recognition accuracy, latency, the system's ability to understand context-specific commands, problems caused by environmental noise, user's accent or speech patterns.

There has been limited research comparing the user performance and user satisfaction of Artificial Intelligence supported voice command interfaces against traditional Virtual Reality controllers. This study aims to compare the two control methods using various metrics like task completion time, participants' exam scores and level of immersion.The hypothesis of this study is that Artificial Intelligence supported voice commands can offer a superior user experience in Virtual Reality gaming by providing a natural form of interaction.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering for the study
* Aged between 20-22 years,
* Being a student in the fourth semester (Spring Semester 2023-2024) of Acibadem Mehmet Ali Aydinlar University Vocational School Anesthesiology Program

Exclusion Criteria:

* No prior Adavanced Cardiac Life Support training,
* History of Virtaul Reality induced motion sickness,
* Medical conditions such as vertigo attacks
* Using medications causing vertigo-like symptoms

Ages: 20 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-07-17 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of two groups' performance scores | Up to 4 weeks
  The participants of two groups will complete a Virtual Reality based exam for performance scoring

SECONDARY OUTCOMES:
Level of immersion during game play | Up to 4 weeks
  The participants of two groups will answer a questionnaire about the level of immersion

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Kitapcioglu, MD, Principal Investigator — Acibadem University
Locations (1):
- Acibadem Mehmet Ali Aydinlar University CASE Simulation Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kitapcioglu D, Aksoy ME, Ozkan AE, Usseli T, Cabuk Colak D, Torun T. Enhancing Immersion in Virtual Reality-Based Advanced Life Support Training: Randomized Controlled Trial. JMIR Serious Games. 2025 Feb 14;13:e68272. doi: 10.2196/68272. PMID 39951703